CLINICAL TRIAL: NCT02147379
Title: Changes in Cognitive Functioning in Euthymic Bipolar Patients Treated With Lurasidone Versus Treatment as Usual; A Randomized, Open-Label Study.
Brief Title: Lurasidone and Cognition in Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H14-00290
Record Dates: First submitted 2014-05-08; First posted 2014-05-26 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Bipolar I Disorder
Keywords: Bipolar Disorder; Cognition; Euthymic; Lurasidone
MeSH Terms: conditions — Bipolar Disorder | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lurasidone (Experimental): Lurasidone 20 - 80 mg / day added to current treatment for 6 weeks.
  Interventions: Drug: Lurasidone
- Treatment as usual (No Intervention): Patients randomized to this arm will continue their usual treatment.

INTERVENTIONS:
Drug: Lurasidone
  Other Names: Latuda
  Arms: Lurasidone

SUMMARY:
This is a 6 week, randomized, open-label, parallel group study in patients with Bipolar-I disorder (manic depression), who are in remission from an episode. Participants who show cognitive impairment at baseline will be randomized to receive open-label Lurasidone added on to their current medication(s) or continue their usual treatment for 6 weeks. Participants will have 3 clinical visits and 2 telephone appointments during the study. Given the preliminary evidence for efficacy of Lurasidone in improving cognition in schizophrenia, we propose to examine the efficacy of Lurasidone in improving cognition in bipolar patients.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must be taking either lithium or valproate or one of the atypical antipsychotics for mood stabilization.
2. Patients who show cognitive impairments (-0.25 standard deviations (SD) or below) on either the Trail Making Test- trial B (TMT-B) or California Verbal Learning Test (CVLT) trials 1 to 5, or CVLT long delay free recall, at baseline visit.
3. Males or females aged 19 to 65 years inclusive.
4. Diagnostic and Statistical Manual IV edition (DSM-IV TR) diagnosis of Bipolar Type I Disorder, with or without a history of psychosis.
5. Clinically stable with a Montgomery Asberg Depression Rating Scale (MADRS) and Young Mania Rating Scale (YMRS) score less than or equal to 8.
6. A sufficient level of English using a language screening questionnaire.
7. Capability of understanding, consenting to, and complying with the requirements of the study.

Exclusion Criteria:

1. A history of unstable or inadequately treated medical illnesses, including moderate to severe brain injury, or neurological illnesses impacting cognitive function.
2. Treatment with Electroconvulsive Therapy (ECT) within eight weeks prior to enrolment; or treatment with an experimental drug within 30 days prior to enrolment.
3. Axis I diagnosis of substance abuse or dependence within the past month.
4. Significant risk of harm to self or others, in the opinion of the investigator.
5. Pregnancy or lactation in female subjects.
6. Liver function tests (AST and ALT) three times the upper limit of normal. -

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-05; Primary Completion 2015-10 (Actual); Study Completion 2017-01-12 (Actual)

PRIMARY OUTCOMES:
Cognitive Change in Bipolar I disorder after treatment with Lurasidone | 6 weeks
  The International Society for Bipolar Disorders-Battery for Assessment of Neurocognition (ISBD-BANC) will be administered to assess cognitive functioning at baseline and at endpoint ( change in scores on cognitive tests) to evaluate the efficacy of lurasidone on cognitive changes in bipolar disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmi N Yatham, MBBS,FRCPC,MRCPsych (UK),MB, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Department of Psychiatry, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Yatham LN, Mackala S, Basivireddy J, Ahn S, Walji N, Hu C, Lam RW, Torres IJ. Lurasidone versus treatment as usual for cognitive impairment in euthymic patients with bipolar I disorder: a randomised, open-label, pilot study. Lancet Psychiatry. 2017 Mar;4(3):208-217. doi: 10.1016/S2215-0366(17)30046-9. Epub 2017 Feb 7. PMID 28185899